CLINICAL TRIAL: NCT05576571
Title: The Utility of Cell-free Methylation Markers in Blood for the Prognosis Prediction of Locoregional Treatment for Hepatocellular Carcinoma
Brief Title: The Utility of Cell-free Methylation Markers in Blood for Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202009079DIPB
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-06

CONDITIONS: Serum Tumor Markers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC case: Patients are those who received radiofrequency ablation or transvascular embolization in National Taiwan University Hospital. Which excludes weakness and inability to cooperate Patients with blood test, under the condition of fully informed consent, complete blood test related tumor indicators (AFP and methylation analysis). The two data are then counted Compare.
  Interventions: Diagnostic Test: Met-score

INTERVENTIONS:
Diagnostic Test: Met-score — methylation analysis

SUMMARY:
Patients with liver cancer expected to undergo radiofrequency ablation or transvascular embolization. Relevant tumor markers (AFP and methylation analysis) were performed. The two data are then counted and compared.

DETAILED DESCRIPTION:
The subjects of this study were patients who were diagnosed with liver cancer by physicians based on AASLD clinical criteria or pathological biopsy.

Patients are those who received radiofrequency ablation or transvascular embolization in National Taiwan University Hospital. Which excludes weakness and inability to cooperate Patients with blood test, under the condition of fully informed consent, complete blood test related tumor indicators (AFP and methylation analysis). The two data are then counted Compare.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with liver cancer by AASLD clinical criteria or pathological sections are planned to receive treatment at National Taiwan University Hospital Liver local treatment such as radiofrequency ablation or transvascular embolization.
2. Be over 20 years old.
3. Under the condition of informed consent, willing to sign the consent form of the subjects.

Exclusion Criteria:

1. Patients who are weak and unable to cooperate with blood test.
2. Kidney dysfunction, serum creatinine greater than 1.5mg/dl, it is judged that computer tomography or MRI cannot be performed Vibrate the injector.

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with liver cancer by AASLD clinical criteria or pathological sections are planned to receive treatment at National Taiwan University Hospital Liver local treatment such as radiofrequency ablation or transvascular embolization.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy (methylation profiling results) | 3 month after treatment
  Correlation of methylation profiling results with AFP and tumor treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD, PhD, Principal Investigator — study principal investigator
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan